CLINICAL TRIAL: NCT01496183
Title: Metabolic Effects of Olanzapine in Healthy Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Steven Dubovsky, principal investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PCH0320106A
Record Dates: First submitted 2011-12-13; First posted 2011-12-21 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Healthy
MeSH Terms: interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Olanzapine (Experimental)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Olanzapine 5mg capsule administered orally at bedtime for 7 days followed by Olanzapine 10 mg capsule administered orally at bedtime for 7 days.
  Arms: Olanzapine
Drug: Placebo — Placebo capsule administered orally at bedtime for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to look at how a two-week use of a medication called Olanzapine might change appetite, physical activity, resting metabolic rate, body composition, and weight in healthy men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer
* Male
* Aged 18-35 years
* Body Mass Index (BMI): <30 kg/m2

Exclusion Criteria:

* Presence of any medical disorder that may confound the assessment of relevant biological measures

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Dubovsky, M.D., Principal Investigator — State University of New York at Buffalo
Locations (1):
- Department of Psychiatry, The State University of New York at Buffalo, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Olanzapine
Started | 9 | 15
Completed | 6 | 13
Not Completed | 3 | 2
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Olanzapine | Total
Number analyzed (Participants) | 6 | 13 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (2.5) | 23.1 (5.1) | 23.6 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 13 | 19
Region of Enrollment [Number; unit: participants]
  United States | 6 | 13 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weight
Time Frame: Assessed at baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: Kg
Groups:
- Placebo: Placebo: Placebo capsule administered orally at bedtime for 14 days Six subjects from the placebo group completed the 2-week double-blind trial and were included in the analysis.
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 6 | 13
Kg | 0.2 (0.5) | 1.7 (1.1)

2. Secondary Outcome: Change From Baseline in Body Composition
Description: lean body mass (kg) and fat mass (kg) at baseline and after 2 weeks of treatment with olanzapine or placebo
Time Frame: baseline and 2 weeks of treatment (olanzapine or placebo)
Population: The Body Composition assessment was not implemented at the start of the study but once the study already started. Therefore, not all study participants who completed the study got the Body Composition assessment done. Only 3 participants in the Placebo Group and 6 participants in the Olanzapine Group got the Body Composition assessment done.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 3 | 6
kg
  lean body mass at baseline | 60.1 (0.7) | 65.8 (11.3)
  lean body mass at 2 weeks of treatment | 60.1 (1.7) | 67.0 (11.7)
  fat mass at baseline | 17.9 (11.7) | 16.5 (9.4)
  fat mass at 2 weeks of treatment | 18.5 (10.0) | 17.4 (8.6)

3. Secondary Outcome: Change From Baseline in 24-Hour Dietary Recall
Description: 24-hour dietary intake recall at baseline and after 2 weeks of treatment with olanzapine or placebo
Time Frame: Assessed at different time points: baseline and 2 weeks of treatment (olanzapine or placebo)
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 6 | 13
kcal/day
  baseline | 1748 (567) | 2410 (1591)
  2 weeks of treatment | 1785 (562) | 2374 (1073)

4. Secondary Outcome: Change From Baseline in Resting Metabolic Rate
Description: Resting metabolic rate at baseline and after 2 weeks of treatment
Time Frame: baseline and 2weeks of treatment
Measure: Mean (Standard Deviation); unit: kcal/24 hours
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 6 | 13
kcal/24 hours
  baseline | 1702 (217) | 1855 (351)
  2 weeks treatment | 1689 (309) | 1858 (342)

5. Secondary Outcome: Change From Baseline Triglycerides
Description: Triglycerides (mg/dl) at baseline and after 2 weeks of treatment with olanzapine or placebo
Time Frame: Assessed at different time points: baseline and 2 weeks of treatment (olanzapine or placebo)
Population: Note regarding the difference between the Overall Number of Participants Analyzed and the Participant Flow: Blood sample could not be collected from 1 participant from the Placebo Group and 1 participant from the Olanzapine Group. Therefore, the number of participants analyzed for the Placebo Group is 5 and for the Olanzapine Group is 12.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 5 | 12
mg/dl
  baseline | 48.4 (13.6) | 93.0 (38.1)
  2 weeks of treatment | 52.8 (22.1) | 136.6 (80.2)

6. Secondary Outcome: Change From Baseline in Glucose
Description: Glucose (mg/dl) at baseline and after 2 weeks of treatment with olanzapine or placebo
Time Frame: Assessed at different time points: baseline and 2 weeks of treatment (olanzapine or placebo)
Population: Note regarding the difference between the Overall Number of Participants Analyzed and the Participant Flow: Blood sample could not be collected from 1 participant from the Placebo Group and 2 participants from the Olanzapine Group. Therefore, the number of participants analyzed for the Placebo Group is 5 and for the Olanzapine Group is 11.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 5 | 11
mg/dl
  baseline | 82.4 (7.4) | 78.6 (8.1)
  2 weeks of treatment | 85.0 (4.2) | 82.2 (5.3)

7. Secondary Outcome: Change From Baseline in Leptin
Description: Leptin (ng/ml) at baseline and after 2 weeks of treatment with olanzapine or placebo
Time Frame: Assessed at different time points: baseline and 2 weeks of treatment (olanzapine or placebo)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 5 | 11
ng/ml
  baseline | 3.8 (3.3) | 3.8 (2.7)
  2 weeks treatment | 4.8 (3.0) | 5.7 (4.3)

8. Secondary Outcome: Change From Baseline in Insulin
Description: Insulin (µIU/ml) at baseline and after 2 weeks of treatment with olanzapine or placebo
Time Frame: Assessed at different time points: baseline and 2 weeks of treatment (olanzapine or placebo)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: µIU/ml
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 5 | 11
µIU/ml
  baseline | 5.0 (3.5) | 6.2 (4.0)
  2 weeks of treatment | 5.8 (2.7) | 10.1 (7.5)

9. Secondary Outcome: Change From Baseline Total Cholesterol
Description: Total cholesterol at baseline and after 2 weeks treatment with olanzapine or placebo
Time Frame: baseline and 2 weeks treatment
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 5 | 12
mg/dl
  baseline | 153.2 (23.7) | 156.8 (32.2)
  2 weeks treatment | 147.4 (21.1) | 167.0 (42.0)

10. Secondary Outcome: LDL
Description: Low-density lipoprotein at baseline and after 2 weeks of treatment with olanzapine or placebo
Time Frame: baseline and 2 weeks treatment
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 5 | 12
mg/dl
  baseline | 88.8 (25.2) | 86.9 (29.2)
  2 weeks treatment | 82.0 (12.5) | 93.7 (34.4)

11. Secondary Outcome: HDL
Description: High-density lipoprotein at baseline and after 2 weeks of treatment with olanzapine or placebo
Time Frame: baseline and 2 weeks treatment
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 5 | 12
mg/dl
  baseline | 54.6 (10.2) | 51.3 (15.7)
  2 weeks treatment | 55.0 (6.8) | 46.1 (11.2)

12. Secondary Outcome: Physical Activity as Measured Using a Physical Activity Monitor
Description: Change from baseline in physical activity. Physical activity was measured using an activity monitor that subjects wore around their waist throughout baseline and treatment days. Subjects were instructed to remove the monitor when sleeping or engaging in water-based activities, and to report on a daily log the times that they were wearing and removing the device. Physical activity was monitored during weekdays and weekend days. Physical activity data were collected in 60-second epochs. The results are reported as average counts per day of physical activity for weekdays and weekend days at baseline and 2 week treatment.
Time Frame: baseline and 2 week treatment
Population: Due to poor participant's compliance with the study requirements for physical activity data collection, the data from 4 participants from the olanzapine group could not be used for analysis purpose.
Measure: Mean (Standard Deviation); unit: counts per day
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 6 | 9
counts per day
  baseline - weekdays | 410,029 (200,091) | 263,720 (131,638)
  2 week treatment - weekdays | 279,722 (119,879) | 263,757 (115,456)
  baseline - weekend days | 279,149 (106,671) | 277,298 (162,147)
  2 week treatment - weekend days | 247,036 (136,553) | 198,382 (117,252)

13. Other Pre Specified Outcome: Laboratory Breakfast Intake
Description: Total kcal intake at breakfast in a laboratory setting at baseline and after 2 week of treatment with olanzapine or placebo
Time Frame: baseline and 2 week treatment
Population: The Laboratory Breakfast Intake assessment was not performed at the start of the study but was initiated during the course of the study. Only 3 participants from the Placebo group and 6 participants from the Olanzapine group completed the Laboratory Breakfast Intake assessment.
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 3 | 6
kcal
  Baseline | 1396 (160) | 864 (269)
  2 week treatment | 1567 (478) | 1058 (482)

ADVERSE EVENTS:
Arm/Group | Placebo | Olanzapine
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/13
Other Adverse Events (participants affected / at risk) | 0/6 | 0/13

LIMITATIONS AND CAVEATS:
The small sample size, the exclusion of obese subjects, and the short olanzapine exposure in the current study may limit the interpretation and generalizability of our findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes